CLINICAL TRIAL: NCT02976077
Title: Preliminary Validation of the RC2S+ Therapy in Schizophrenia
Brief Title: RC2S+: Remediation of Social Cognitive Impairments
Acronym: RC2S+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-A01271-50
Record Dates: First submitted 2016-11-16; First posted 2016-11-29 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Schizophrenia
Keywords: social cognition; cognitive remediation; emotions; theory of mind; attributions; social perception
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- RC2S+ (Experimental): RC2S+
  Preparation sessions (sessions 1 & 2):
  * Functional Outcomes Scale - Social Cognition (ERF-CS)
  * Psychoeducation about social cognitive impairments
  * Concrete objectives
  Cognitive remediation (sessions 3 to 22):
  * Paper-and-pencil session
  * Simulation session
  * Home-based task
  Transfer sessions (sessions 23 & 24):
  * Transfer of skills in dayly life - generalization
  * Assessment of the achievement of objectives
  Interventions: Behavioral: RC2S+
- Control therapy (Active Comparator): Control therapy
  Preparation sessions (sessions 1 & 2):
  * Functional Outcomes Scale - Neurocognition
  * Psychoeducation about cognitive impairments
  * Concrete objectives
  Cognitive remediation (sessions 3 to 24):
  * Paper-and-pencil session
  * Simulation session
  * Home-based task
  Interventions: Behavioral: active comparator

INTERVENTIONS:
Behavioral: RC2S+ — new cognitive remediation program
  Arms: RC2S+
Behavioral: active comparator — cognitive remediation program
  Arms: Control therapy

SUMMARY:
Background:

Difficulties in social interactions are a central characteristic of people with schizophrenia, and can be partly explained by impairments of social cognitive processes. According to renown researchers, three to five social cognitive processes are usually altered in schizophrenia: (1) emotional processing; (2) theory of mind (ToM); (3) attributional style; and (4 and 5) social perception and knowledge. The components of social cognition appear to be related to both symptomatology and functioning in everyday life.

New strategies of cognitive remediation have been recently developed to target these deficits and few meta analyses have assessed the extent to which social cognitive remediation programs have led to multiple improvements for schizophrenia patients. Overall, it seems that such therapies showed encouraging results in both patient interest and motivation, and social cognitive processes.

The RC2S therapy is the first individualized and partly computerized program through which patients practice social interactions and develop social cognitive abilities with simulation techniques in a realistic environment.

DETAILED DESCRIPTION:
Methods:

This is a randomized controlled trial to establish the validity of the RC2S+ program in schizophrenia.

The project's main objective is to assess the impact of RC2S+ on social cognitive impairments in schizophrenia compared with a cognitive remediation program (control therapy) focusing on neurocognition, equivalent in terms of number, duration and rhythm of sessions.

The study has four other objectives:

1. To assess the influence of the RC2S+ therapy versus control therapy on neurocognitive processes
2. To assess the impact of the RC2S+ therapy versus control therapy on social functioning
3. To assess the impact of the RC2S+ therapy versus control therapy on both positive and negative symptoms
4. To study the maintenance of benefits 3 months forward

Outcomes:

To treat social cognitive impairments in people with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years old
* Diagnosis of schizophrenia assessed with DSM5 criteria (APA, 2013)
* No modification of psychotropic treatment during the month before inclusion (variation of 20% of the dose is tolerated
* French native language or education in a French school since the first year of primary school
* Consent to participate to the study and agreement of the legal guardian
* Patients who have not benefited from cognitive remediation during the three months before inclusion

Exclusion Criteria:

* Substance use disorder (criteria of DSM-5), except for caffeine and tobacco
* Neurologic disorders (vascular, infectious or neurodegenerative)
* Uncorrected visual deficit
* Medical drugs with cerebral or psychological effect (e.g, corticosteroids)
* Patients resistant to antipsychotic medication
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the HB (Hostility Bias) score | week 12
  AIHQ (Ambiguous Intentions Hostility Questionnaire)

SECONDARY OUTCOMES:
Change from baseline in social cognitive | week 12
  ACSO ( Self-Assessment Scale of Social Cognition Disorders)
Change from baseline in episodic verbal learning and memory | week 12
  CVLT( California Verbal Learning Test),
Change from baseline in visual attention and task switching | week 12
  TMT( Trial Making Test)
Change from baseline in social functioning | week 12
  FEFSF (First Episode Social Functioning Scale)
Change from baseline in symptoms at week 12 | week 12
  PANSS (Positive And Negative Symptoms Scale)
Change from baseline in visuospatial abilities at week 12 | week 12
  TMT( Trial making Test)
Change from baseline in executive functioning at week 12 | week 12
  FNART(French National Adult reading Test)

CONTACTS AND LOCATIONS:
Overall Officials: FRANCK NICOLAS, PUPH, Principal Investigator — LE VINATIER HOSPITAL BRON FRANCE
Locations (1):
- centre de réhabilitation - Hôpital le Vinatier, Lyon, Rhône, France

REFERENCES:
- [Derived] Peyroux E, Prost Z, Amado I, Graux J, Demily C, Plasse J, Franck N; RC2S Consortium. Is the Cognitive Remediation of Social Cognition (RC2S) program useful to improve social cognition and functional outcomes in people with schizophrenia? A randomized controlled trial. Psychiatr Rehabil J. 2026 Jan 12. doi: 10.1037/prj0000673. Online ahead of print. PMID 41525374